CLINICAL TRIAL: NCT02479360
Title: A Study Investigating the Inter- and Intra- Rater Reliability of a Battery of Functional Standardised Outcome Measures in Neurofibromatosis 1
Brief Title: Reliability of Functional Outcome Measures in Neurofibromatosis 1
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RJ115/N174
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-06

CONDITIONS: Neurofibromatosis 1, NF1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outcome measurement: Each participant will be asked to complete each standardised outcome measure (SOM) three times and each trial will be videotaped by the researcher. The selected SOM's are the 10 metre walk test, the timed up and go test, the functional reach test and the nine-hole peg test. A physiotherapist will watch the video on 2 separate occasions to evaluate intra-rater reliability. Inter-rater reliability will be assessed through asking three other neurofibromatosis specialist professionals (two NF1 consultants and one NF1 specialist nurse) to review the video and to score each measure completed. Once the filmed sessions have been analysed by the relevant clinician's the data will be destroyed in line with Trust policy.

SUMMARY:
Neurofibromatosis 1 (NF1) is a common inherited condition that affects the skin, bone and nervous system. The complications of NF1 are widespread and can lead to varied difficulties dependent on the location of neurofibromas and their secondary complications. At present evaluation of the effect of treatments in NF1 is based on a clinician's neurological assessment, magnetic resonance imaging and positron emission tomography but it is apparent that imaging results do not always link with clinical and functional changes in an individual. This study aims to evaluate the reliability (stability) of a range of functional standardised outcome measures in adults with NF1.

DETAILED DESCRIPTION:
Neurofibromatosis 1 (NF1) is an inherited condition that occurs in 1 in 2,500 births; affecting the skin, bone and nervous system. The complications of NF1 are widespread and can lead to varied difficulties dependent on the location of neurofibromas and their secondary complications. One person with NF1 may have minimal issues whereas another may be profoundly disabled; one may have difficulties using their hands and arms and another may have difficulties standing from a chair. New pharmacological and nonpharmacological treatments for NF1 are currently being developed and they have potential to dramatically influence a person with NF1's life. At present evaluation of treatment effect in NF1 is based on a clinician's neurological assessment, magnetic resonance imaging and positron emission tomography and it is apparent that imaging results do not always link with clinical and functional changes in an individual. Therefore clinicians and researchers agree that the analysis of treatment effect needs to include the evaluation of a person's function. The findings from this study will improve the care of people with NF1 by ensuring that we are able to measure functional changes in a person with NF1 with greater confidence, meaning that we can start, continue or cease treatments based on the holistic picture of an individual.

The world confederation of physiotherapists (WCPT) stipulates that standardised outcome measures (SOM) are used to provide a quantitative measure of capability, and to evaluate the impact of treatment on function. There are a wide range of SOM's that evaluate function (e.g. walking, standing from a chair, use of hands) so a SOM is chosen by the clinician based on the patient's presenting functional difficulty and the scientific credibility of the SOM. Scientific credibility (robustness) is based on scientific properties of the SOM i.e. how stable the SOM is (reliability) and whether it assesses what it is intending to assess (validity). It is important to evaluate each SOM within the target population as variability within that condition, strongly influences the SOM's reliability and validity (de Vel 2011).

At present, functional SOM's have limited scientific and subsequent clinical credibility when used in people with NF1 because their scientific properties have not yet been evaluated within this patient group which means that if they are used clinically or within research, there is an inherent element of doubt when interpreting the SOM's results. The objective of this research team is to create a core set of functional SOM's which have undergone rigorous scientific evaluation so that they can be used in the future for clinical practice and for research purposes in adults with NF1.

This study aims to evaluate four commonly used SOM's for reliability in adults with NF1 (over 16 years of age). The measures chosen for evaluation are the 10 metre walk test, the timed up and go test, the functional reach test and the nine hole peg test. Interrater reliability (the test result remains the same when reviewed by different people) and intrarater reliability (the test result remains stable when reviewed twice by the same tester) will be evaluated. From this data, we will be able to calculate the standard error of measurement an additional important scientific characteristics of SOM evaluation.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 16 years or older who fulfil the diagnostic criteria for NF1 who do not have a significant mobility or balance impairment that is unrelated to their NF1,
* Able to walk more than 10 metres without physical assistance (may use walking aids)
* Patients who attend the national NF1 service at GSTT

Exclusion Criteria:

* Patients who are unable to provide informed consent will be unable to participate in this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adults (over the age of 16 years) with a clinical diagnosis of neurofibromatosis 1 who attend the neurofibromatosis clinic for appointments at Guys hospital, London and who fit the inclusion/exclusion criteria for the trial are eligable to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
10 metre walk test | Between 5 and 30 seconds per test on average.
  Participant is asked to stand at a point 2.5m before the start of a 10 metre walk way. They are advised to walk at their 'normal speed' from here to (a point 2.5m beyond the 10m walk way). The assessor times from the moment the participant's leading foot crosses the start point for the 10 metre walk way until the toes of the participant's leading foot crosses the end of the 10m walk way. Measurements are recorded in seconds and milliseconds. Participants can use their normal aids and orthotics if needed.
Functional Reach test | 30 seconds per test
  Participant stands with arms straight out in front of him/herself at shoulder level and hands forming fists. The assessor sticks a ruler to the wall at the end of their hands. Participant is advised to lean forwards as far as they can without falling over and the assessor measures the distance they can reach against the metre ruler in centimetres and millimetres.
9 hole peg test | Up to 60 seconds per hand.
  Participant is sitting comfortably in a chair in front of a desk. The 9 hole peg test equipment is set up so that the bowl containing pegs is directly behind the pegboard and in front of the participant. Participants can rest the forearms on the desk but must use only 1 hand for each test. If not the test is invalid. The assessor measures from the time the fingers pick up the first peg from the bowl until the fingers place the last peg in the hole of the pegboard. Time will be recorded in seconds and milliseconds.
Timed up and go test | Up to 60 seconds
  Participant sits in a chair at the end of the 3m walkway. S/he is asked to stand up from the chair walk to the line, turn around once they reach the line and return to the chair. If they do not touch the line during the test, the test is invalid. The participant can use any aids/ orthotics that they normally use. The assessor will time from the moment the participants back leaves the backrest until it touches it again at the end of the test. Time will be recorded in seconds and milliseconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurofibromatosis Unit, Guys Hospital., London, United Kingdom